CLINICAL TRIAL: NCT03746080
Title: A Follow-Up Study to Add Whole Brain Radiotherapy (WBRT) to Standard Temozolomide Chemo-Radiotherapy in Newly Diagnosed Glioblastoma (GBM) Treated With 4 Weeks of Continuous Infusion Plerixafor
Brief Title: Whole Brain Radiation Therapy With Standard Temozolomide Chemo-Radiotherapy and Plerixafor in Treating Patients With Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lawrence D Recht (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Lawrence D Recht, Professor of Neurology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-46410; NCI-2018-02159 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BRN0037 (Other: OnCore Number); IRB-46410 (Other: Stanford IRB)
Record Dates: First submitted 2018-11-07; First posted 2018-11-19 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma; Glioblastoma With Primitive Neuronal Component; Gliosarcoma; Malignant Glioma; Oligodendroglial Component Present
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Glioma | interventions — plerixafor; ferric pyrophosphate; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Whole Brain Radiotherapy + Plerixafor +Chemoradiotherapy (Experimental): After completion maximal safe surgical resection, patients undergo radiation therapy for 42 days, initiating whole brain radiation therapy at day 21 (dose 16 of radiation therapy) and receive temozolomide daily on days 1 to 42. Beginning 7 days before the completion of whole brain radiation therapy, patients receive plerixafor by continuous infusion on days to 1 to 28. Beginning 1 week after completion of plerixafor infusion and 35 days after completion of whole brain radiation therapy, patients receive temozolomide monthly for 6 to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Plerixafor; Drug: Temozolomide; Radiation: Whole-Brain Radiotherapy (WBRT); Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Plerixafor — Plerixafor will be administered via infusion at 400 micrograms per kilogram per day for four weeks beginning one week before the end of radiation
  Other Names: AMD 3100; JM-3100; Mozobil; SDZ SID 791
Drug: Temozolomide — Temozolomide (TMZ) will be administered concurrently with the radiation for 42 days and 6-12 cycles of monthly adjuvant Temozolomide (TMZ) after completion of Plerixafor infusion.
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac
Radiation: Whole-Brain Radiotherapy (WBRT) — Undergo Whole brain radiotherapy (WBRT) - Radiotherapy consists of 30 Gy in 15 fractions of whole brain radiations
  Other Names: WBRT; whole-brain radiation therapy; whole-brain radiotherapy
Radiation: Radiation Therapy — Radiotherapy consists of 30 Gy in 15 fractions
  Other Names: XRT; RT

SUMMARY:
This phase II trial studies how well whole brain radiation therapy works with standard temozolomide chemo-radiotherapy and plerixafor in treating patients with glioblastoma (brain tumor). Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Plerixafor is a drug that may prevent recurrence of glioblastoma after radiation treatment. Giving whole brain radiation therapy with standard temozolomide chemo-radiotherapy and plerixafor may work better in treating patients with glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary purpose of this Phase II study is to evaluate the efficacy of Plerixafor administered with a modified radiation regimen that includes a component of WBRT. The primary endpoint is 6-month progression free survival post initiation of Chemoradiation.

SECONDARY OBJECTIVES:

I. To assess the median survival of patients treated with continuous infusion plerixafor/WBRT.

II. To assess the toxicities both short and long term of continuous infusion plerixafor/WBRT.

III. To assess the patterns of failure (in and out of irradiated brain field, out of brain) of continuous infusion plerixafor/WBRT.

OUTLINE:

After completion maximal safe surgical resection, patients undergo radiation therapy for 42 days, initiating whole brain radiation therapy at day 21 (dose 16 of radiation therapy) and receive temozolomide daily on days 1-42. Beginning 7 days before the completion of whole brain radiation therapy, patients receive plerixafor by continuous infusion on days 1-28. Beginning 1 week after completion of plerixafor infusion and 35 days after completion of whole brain radiation therapy, patients receive temozolomide monthly for 6-12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for adverse events for 30 days after the last dose of Plerixafor and then every 12 weeks for 5 years for survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have tissue confirmation of high grade (World Health Organization (WHO) grade IV) glioma including but not limited to glioblastoma, gliosarcoma, glioblastoma with oligodendroglial features, glioblastoma with primitive neuroectodermal tumor (PNET) features.
* The patient must have post-operative contrast enhanced imaging (computed tomography [CT] or magnetic resonance imaging [MRI]) unless only biopsy performed. For patients having biopsy alone, post-operative imaging is not routinely obtained and therefore the preoperative study will serve as baseline.
* Patient should have surgery (biopsy, partial resection or gross total resection) and no additional anti-cancer therapy except the chemo-radiation as specified in the protocol.
* Patients must have Karnofsky performance score >= 60.
* Absolute neutrophil count (ANC) >= 1500 (at time of screening).
* Platelets >= 100,000 ml (at time of screening).
* Serum creatinine =< 1.5mg/dl (at time of screening).
* Creatinine (Cr) clearance should be > 50 mL/min (at time of screening).
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 times the upper limit of normal (at time of screening).
* If female of childbearing potential, negative pregnancy test (at time of screening).
* The patient or his/her legal representative must have the ability to understand and willingness to sign a written informed consent document.
* Patient agrees to use an effective method of contraception (hormonal or two barrier methods) while on study and for at least 3 months following the plerixafor infusion.

Exclusion Criteria:

* Prior or concurrent treatment with Avastin (bevacizumab).
* Prior exposure to plerixafor.
* Prior use of other investigational agents to treat the brain tumor.
* Recent history of myocardial infarct (less than 3 months) or history of active angina.
* Prior malignancy except for non-melanoma skin cancer and carcinoma in situ (of the cervix or bladder), unless diagnosed and definitively treated more than 3 years prior to 1st dose of investigational drug.
* Prior sensitivity to plerixafor.
* Pregnant or patients who are breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2024-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Recht, Principal Investigator — Stanford Cancer Institute Palo Alto
Locations (1):
- Stanford Cancer Institute Palo Alto, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 21 participants signed informed consent; 17 participants were allocated to treatment; 2 patients still in follow up
Period: Overall Study
Arm/Group | Whole Brain Radiotherapy + Plerixafor +Chemoradiotherapy
Started | 17
On treatment | 17
Completed treatment | 17
Completed | 0
Not Completed | 17
Not completed — In follow up | 2
Not completed — Death | 15

BASELINE CHARACTERISTICS:
Arm/Group | Whole Brain Radiotherapy + Plerixafor +Chemoradiotherapy
Number analyzed (Participants) | 17
Age, Customized [Count of Participants; unit: Participants]
  18 to 30 years | 1
  31 to 39 years | 1
  40 to 49 years | 3
  50 to 59 years | 6
  60 to 69 years | 4
  70 to 79 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Progression Free Survival Participants (PFS) at Six Months
Description: Proportion of Progression free survival will be measured at 6 months post initiation of chemoradiation. Simon 2-stage design will be use to assess progression-free survival. Will be computed from start of induction therapy and summarized with Kaplan-Meier estimates.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Whole Brain Radiotherapy + Plerixafor +Chemoradiotherapy
Number analyzed (Participants) | 17
Proportion of participants | 0.786 [0.598 to 1.0]

2. Secondary Outcome: Median Survival
Description: Median survival will be assessed at 31 months of subjects who have completed the 28 day Plerixafor infusion. Will be computed from start of induction therapy and summarized with Kaplan-Meier estimates.
Time Frame: up to 31 months
Measure: Median (Standard Error); unit: days
Arm/Group | Whole Brain Radiotherapy + Plerixafor +Chemoradiotherapy
Number analyzed (Participants) | 17
days | 398 (0.134)

3. Secondary Outcome: Toxicity Associated With Plerixafor/WBRT
Description: Incidence of adverse events will be graded and recorded per Common Terminology Criteria for Adverse Events version 5.0. Will assess reported toxicities up until 30 days of treatment. The number of participants experiencing adverse events, including qualifying dose limiting toxicities (DLTs) will be tabulated by attribution (Unrelated, Unlikely to be related, Definitely related) and severity.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Brain Radiotherapy + Plerixafor +Chemoradiotherapy
Number analyzed (Participants) | 17
Participants
  Grade 3 or higher AE | 3
  Related to WBRT treatment | 1
  Related to Plerixafor treatment | 0

4. Secondary Outcome: Patterns of Treatment Failure
Description: Patterns of Failure in patients receiving Whole Brain Radiotherapy + Plerixafor + Chemoradiotherapy was assessed by determining the out-of-field occurrence or occurrence outside of the brain over time. Local treatment failure was defined as within the 95% isodose region. Out-of-field occurrence is defined by any treatment failure observed outside treatment area.
Time Frame: 5 years
Population: Participants with available scan data were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Whole Brain Radiotherapy + Plerixafor +Chemoradiotherapy
Number analyzed (Participants) | 14
Participants
  In Field Occurrence | 12
  Out-of-field Occurrence | 2

ADVERSE EVENTS:
Time Frame: All-Cause Mortality monitored/assessed up to 31 months. Serious and Other (Not Including Serious) Adverse Events were monitored/assessed 30 days after the completion of 28-day Plerixafor infusion.
Arm/Group | Whole Brain Radiotherapy + Plerixafor +Chemoradiotherapy
All-Cause Mortality (participants affected / at risk) | 15/17
Serious Adverse Events (participants affected / at risk) | 3/17
Other Adverse Events (participants affected / at risk) | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Whole Brain Radiotherapy + Plerixafor +Chemoradiotherapy (N=17)
Depression (Psychiatric disorders) | 1 (1)
Cerebral Edema (Nervous system disorders) | 1 (1)
Pseudo Progession (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Whole Brain Radiotherapy + Plerixafor +Chemoradiotherapy (N=17)
Anemia (Blood and Lymphatic System Disorders) | 1 (1)
Palpitations (Cardiac Disorders) | 1 (1)
Supraventricular Tachycardia (Cardiac Disorders) | 1 (1)
Tinnitus (Ear and Labyrinth Disorders) | 1 (1)
Hearing Impaired (Ear and Labyrinth Disorders) | 1 (1)
Floaters (Eye Disorders) | 1 (2)
Excessive Eye discharge/Rheum (Eye Disorders) | 1 (1)
Eye Irritation (Eye Disorders) | 1 (1)
Abdominal Pain (Gastrointestinal Disorders) | 1 (1)
Constipation (Gastrointestinal Disorders) | 4 (4)
Diarrhea (Gastrointestinal Disorders) | 5 (5)
Dyspepsia (Gastrointestinal Disorders) | 2 (2)
Hypersalivation (Gastrointestinal Disorders) | 1 (1)
Nausea (Gastrointestinal Disorders) | 12 (14)
Toothache (Gastrointestinal Disorders) | 1 (1)
Vomiting (Gastrointestinal Disorders) | 6 (12)
Chills (General Disorders) | 3 (3)
Edema face (General Disorders) | 1 (1)
Fatigue (General Disorders) | 11 (12)
Lump on the back of neck (General Disorders) | 1 (1)
Gait disturbance (General Disorders) | 1 (2)
Non-cardiac chest pain (General Disorders) | 1 (1)
Pain (General Disorders) | 1 (1)
Conjunctivitis (Infections and Infestations) | 2 (2)
Shingles (Infections and Infestations) | 1 (1)
Thrush (Infections and Infestations) | 1 (1)
Dermatitis radiation (Injury, Poisoning and procedural complications) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 6 (7)
Platelet count decreased (Investigations) | 4 (6)
Anorexia (Metabolism and Nutrition Disorders) | 3 (3)
Hypokalemia (Metabolism and Nutrition Disorders) | 1 (1)
Hyponatremia (Metabolism and Nutrition Disorders) | 2 (2)
Neck Pain (Musculoskeletal and Connective Tissue Disorders) | 1 (1)
Muscle cramp (Musculoskeletal and Connective Tissue Disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and Connective Tissue Disorders) | 2 (2)
Pain in extremity (Musculoskeletal and Connective Tissue Disorders) | 1 (1)
Back pain (Musculoskeletal and Connective Tissue Disorders) | 1 (1)
Pain in extremity R foot (Musculoskeletal and Connective Tissue Disorders) | 1 (1)
Anosmia (Nervous System Disorders) | 2 (2)
Ataxia (Nervous System Disorders) | 1 (1)
Cognitive disturbance (Nervous System Disorders) | 3 (3)
Dizziness (Nervous System Disorders) | 4 (4)
Dysgeusia (Nervous System Disorders) | 2 (3)
Headache (Nervous System Disorders) | 5 (7)
Lethargy (Nervous System Disorders) | 1 (1)
Memory Impairment (Nervous System Disorders) | 1 (1)
Imbalance (Nervous System Disorders) | 2 (2)
Muscle weakness left-sided (Nervous System Disorders) | 1 (1)
Muscle weakness, lower limb (Nervous System Disorders) | 1 (1)
Paresthesia (Nervous System Disorders) | 2 (2)
Presyncope (Nervous System Disorders) | 1 (1)
Somnolence (Nervous System Disorders) | 1 (1)
Tremor (Nervous System Disorders) | 2 (2)
Visual field disturbance (Nervous System Disorders) | 1 (1)
Right hand focal motor movement (Nervous System Disorders) | 1 (1)
Confusion (Psychiatric Disorders) | 1 (1)
Agitation (Psychiatric Disorders) | 1 (1)
Delirium (Psychiatric Disorders) | 2 (2)
Depression (Psychiatric Disorders) | 1 (1)
Insomnia (Psychiatric Disorders) | 4 (4)
Irritability (Psychiatric Disorders) | 1 (1)
Labile mood (Psychiatric Disorders) | 1 (1)
Suicidal ideation (Psychiatric Disorders) | 2 (2)
Anxiety (Psychiatric Disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Cough (Respiratory, Thoracic and Mediastinal Disorders) | 1 (1)
Dyspnea (Respiratory, Thoracic and Mediastinal Disorders) | 1 (1)
Allergic Rhinitis (Respiratory, Thoracic and Mediastinal Disorders) | 1 (1)
Epistaxis (Respiratory, Thoracic and Mediastinal Disorders) | 1 (1)
Sore throat (Respiratory, Thoracic and Mediastinal Disorders) | 1 (1)
Flushing (Vascular Disorders) | 1 (1)
Hot flashes (Vascular Disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT03746080/Prot_SAP_000.pdf